CLINICAL TRIAL: NCT03171376
Title: Effect of Coronal Extent of Obturation in Relation to Marginal Bone on Endodontic - Periodontal Lesions Without Communication: A Randomized Controlled Trial
Brief Title: Effect of Coronal Extent of Obturation on Endo-perio Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Gaurav
Record Dates: First submitted 2017-05-24; First posted 2017-05-31 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2017-09

CONDITIONS: Apical Periodontitis
Keywords: Root canal treatment; Coronal leakage; Intraorifice barrier
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intraorifice Group (Active Comparator): After root canal treatment intraorifice barrier of glass-ionomer cement (Ketac™ Molar, 3M ESPE ) placed 3mm inside canals from root canal orifice.
  Interventions: Procedure: Root canal treatment and coronal restoration
- Base Group (Active Comparator): 2mm thick base of glass-ionomer cement (Ketac™ Molar, 3M ESPE ) applied uniformly on the floor of the pulp chamber after completion root canal treatment.
  Interventions: Procedure: Root canal treatment and coronal restoration
- Control Group (Active Comparator): Neither intraorifice barrier nor base applied after completion of root canal treatment.
  Interventions: Procedure: Root canal treatment and coronal restoration

INTERVENTIONS:
Procedure: Root canal treatment and coronal restoration — After primary root canal treatment, Glass Ionomer Cement (Ketac™ Molar, 3M ESPE) applied as intraorifice barrier 3mm inside canal from root canal orifice in first group, as 2mm base on floor of pulp chamber in second group and direct composite restoration in 3rd group without Intraorifice barrier or base.

SUMMARY:
Increased incidence of apical periodontitis was reported where root filling was found coronal to the marginal bone due to communication between pulp and periodontal space. It has been suggested to place intraorifice barrier in the canal to provide coronal seal. However there exists a void in literature regarding clinical validity of the termination of obturation apical to marginal bone and placement of intraorifice barrier in resolution of periapical pathology. Therefore this randomized controlled trial intends to investigate effect of coronal level of obturation on endodontic success and marginal breakdown.

DETAILED DESCRIPTION:
TITLE : " Effect of coronal extent of obturation in relation to marginal bone on the healing of endodontic - periodontal lesions without communication: a randomized controlled trial."

INTRODUCTION: Coronal leakage is considered significant factor for failure of endodontic treatment . To provide endodontic care of highest quality attention should be given to coronal restoration after successful completion of root canal treatment. In an array of retrospective studies significant numbers of cases were reported of apical periodontitis in teeth with unsatisfactory coronal seal as compared to the ones with clinically or radiographically acceptable coronal restoration. Post treatment restorative status and quality & extent of root filling along with preoperative periapical lesion were found to have strong effect on outcome of endodontic treatment.

Gutta-percha and sealer alone used routinely as root canal obturating material are found to be ineffective to guard against microleakage. Even clinically acceptable root filling allow penetration of bacteria and their products in as less as three days and contribute to eventual treatment failure. This breach of seal in coronal segment of obturated root canal may significantly jeopardize endodontic treatment outcome particularly in molars because of presence of accessory canals in the floor of the pulp chamber.

Placing an additional protective barrier in the coronal portion of the root canal has been recommended to minimize microleakage and facilitate healing of apical periodontitis. Intraorifice barrier apart from enhancing probability of success of endodontic treatment may also augment periodontal therapy as intra pulpal infection is known to contribute in worsening of periodontal health by promoting marginal bone loss and pocket formation.

Many materials have been tried as intraorifice barrier like cavit, IRM, amalgam, GIC, composite resin, dentin bonding agents, MTA. Some studies have reported no difference amongst materials while other found better performance of MTA over composite/GIC ; GIC over Polycarboxylate cement/Flowable composite and resilon alone without intraorifice barrier and composite over MTA/Cavit12 and Cavit/IRM.Recent studies have advocated use of adhesive restorative material like GIC to provide adequate seal against bacterial micro leakage. Lee et al demonstrated better sealing ability of MTA over both composite and GIC in an in vitro dye infiltration experiment. Glass ionomer may provide better seal against penetration of bacteria to the periapex because of its adhesive nature and ability to bond to the sclerotic dentin found on the pulpal floor better than composite resin.

However concerns are raised while applying these results in clinical setting because of varied methodology employed in these studies. Also in a review article Gillen et al pointed out that coronal restoration may be overemphasised based on the results of the in vitro studies. So It remain to be seen whether the success of intraorifice barrier in preventing microleakage is translated from in vitro studies in to the clinical setting which by far is more challenging, variable and difficult to interpret.

Few animal studies have compared the efficacy of coronal plug in preventing periapical inflammation. Animal studies in dog have reported minimal or no periapical inflammation in teeth with MTA intraorifice barrier than the ones without intraorifice barrier. Stassen et al in an retrospective study evaluated the effect of intraorifice barrier in relation to marginal bone level and found more cases of apical periodontitis in tooth where root filling extended coronal to marginal bone level called positive than the ones where the root filling ended apical to marginal bone level called negative on the healing of apical periodontitis. While depth of intraorifice barrier has been investigated earlier. Level of intraorifice barrier and its effect on propagation of marginal periodontitis and healing of apical periodontitis remain unexplored.

So far no prospective clinical trial has investigated the effect of intraorifice barrier on the healing of marginal and apical periodontitis after successful root canal treatment. In absence of a clinical study substantial amount of doubt still persists whether intraorifice barrier can emerge as an effective mean to prevent microleakage in furcation and root canals of a multirooted tooth which because of its anatomical aberrations poses stiff challenge for clinicians.

Therefore aim of this randomised controlled trial is to determine effect of the coronal extent of obturation in relation to marginal bone on the marginal breakdown and periapical healing and to determine effect of intracanal glass ionomer restoration as intraorifice barrier on treatment outcome of apical periodontitis.

AIMS AND OBJECTIVES

1. To determine effect of the coronal extent of obturation in relation to marginal bone on the marginal breakdown and periapical healing.
2. To determine effect of intracanal glass ionomer restoration as intraorifice barrier on treatment outcome of apical periodontitis.

MATERIALS AND METHODOLOGY

This study is conducted in the department of conservative dentistry and endodontics, post graduate institute of dental sciences, Rohtak. Study subjects were obtained from the pool of OPD patients in the Department of conservative dentistry and endodontics, PGIDS, Rohtak.

METHODOLOGY Prior to treatment a thorough clinical and radiological examination was carried out.

A thorough history was taken from each patient. Prior informed consent was taken after explaining the procedure, risks and benefits.

Clinical procedure:

A total of 60 patients (n=20 in each group) were included in the study.

Sample size determination:

Sample of 16 patients each was calculated based on the difference in periapical inflammation with and without intraorifice barrier(39% and 89% respectively) in an animal study conducted by Yamauchi et al.

Considering the attrition rate of 25% sample of 20 patients each were recruited in the study.

Mature mandibular permanent molar with diagnosis of apical periodontitis (as confirmed clinically & by periapical radiograph) were chosen for the study.

All periapical radiographs were exposed by using constant kVP, mA and exposure time (70 KVP, 8 mA, 0.8 sec.) After initial periodontal therapy, administration of local anesthesia, rubber dam isolation of the involved tooth was done.

Caries excavation was done and access cavity was prepared using carbide burs in high speed handpiece with copious irrigation.

Debridement of the pulp chamber was done and all canal orifices were identified.

Negotiation of canals was done. Working length was determined using root ZX apex locator and were verified radiographically.

After creating glide path with #15 k-file, Revo-S (Micro Mega, Besancon, France) instruments were used in sequence as suggested by manufacturer recommendation with a rotational speed of 350 rpm in gentle in-out motion. The torque was adjusted to 2.5 Ncm, and a crown-down approach was selected. Once, the instrument had negotiated to the end of the canal and had rotated freely, it was removed.

Irrigation was carried out using 5 mL of a 5.25% NaOCl solution between files. After preparation, the root canals were irrigated with 5 mL 17% EDTA for 3 minutes to remove smear layer, followed by 5 mL 5.25% NaOCl. The final irrigation was done with 5 mL distilled water.

The root canals was dried using paper points and filled with laterally condensed gutta-percha (Meta Biomed Co Ltd, Korea) and Roth R-801 sealer (Roth International Drug Co., Chicago, Ill) mixed according to manufacturers' instructions.

Gutta-percha was cut with a heated instrument and vertically condensed right at the orifice opening of the canals.

The teeth were randomly divided into 3 experimental groups of 20 teeth each as follows :

1. Group I: intraorifice barrier of glass-ionomer cement (Ketac™ Molar, 3M ESPE) placed 3mm in the canal from root canal orifice.
2. Group II: base of 2mm of glass-ionomer cement (Ketac™ Molar, 3M ESPE) placed on the floor of the pulp chamber.
3. Group III: control group with neither intraorifice barrier placed nor base applied.

Method of randomization Using an equal proportion randomization allocation ratio, one of the investigators created envelopes containing concealed assignment codes that was assigned sequentially to eligible patients. It was ensured that neither the investigator nor the patient were aware of the treatment protocol at the time of patient allocation.

Glass Ionomer Cement (Ketac™ Molar, 3M ESPE) was mixed according to manufacturer's instructions.

In group I: The gutta-percha was removed 3mm from the coronal portion of the canal with hot plugger. Excess root canal sealer was removed with sterilized alcohol-wet cotton pellets. Glass Ionomer Cement was applied inside canal and condensed as well as 2mm thick uniform base on the floor of the pulp chamber.

In group II 2mm thick base of Glass Ionomer Cement was applied uniformly on the floor of the pulp chamber with plastic instrument.

Final composite restoration was placed in all groups according to the manufacturer's instruction.

Periodontal therapy in the form of scaling and root planning was done on the day endodontic treatment completed.

FOLLOW UP Follow up and clinical and radiographic examination is carried out at 3, 6, 9 & 12 month period.

ELIGIBILITY:
Inclusion Criteria:

1. Mature permanent mandibular molars.
2. Pulpal necrosis as confirmed by negative response to pulp sensibility test (cold and electric pulp test) ;
3. Radiographic evidence of apical periodontitis in the form of periapical radiolucency (size not more than 2 × 2 mm);
4. Generalized chronic periodontitis criteria will be considered when ≥ 30% of sites will be involved with clinical attachment loss (CAL) slight = 1or 2mm, Moderate = 3-4mm, and severe ≥ 5mm.
5. Probing depth<4mm
6. Radiographic alveolar bone breakdown not more than one third of root length.

Exclusion Criteria:

1. Younger than 18 years;
2. Pregnant, diabetic, or immunocompromised;
3. Having a positive history of antibiotic use within the past month or require antibiotic premedication for dental treatment (including infective endocarditis or prosthetic joint prophylaxis);
4. Teeth having previous root fillings, unrestorable teeth, fractured/perforated roots, grade 3 mobility, and history of recent periodontal therapy (within previous 6 months); and
5. Teeth with established endodontic-periodontal lesions exhibiting <2 mm radiopaque bone between the root apex.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Clinical success | Baseline to one year.
  Success was defined as absence of signs and symptoms and reduction in pocket depth measured in millimeter.
Radiographic Success | Baseline to one year
  Absence of periapical alterations (radiolucency at furcal or periapical region).

IPD SHARING:
Plan to Share IPD: Yes